CLINICAL TRIAL: NCT01976689
Title: New- Onset Diabetes and Glucose Regulation Are Significant Determinants of Left Ventricular Hypertrophy in Renal Transplant Recipients
Brief Title: New-onset Diabetes and Left Ventricular Hypertrophy in Renal Transplantation
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Mehtap Erkmen Uyar, Md, Neprology Fellow, Baskent University
Other Study IDs: TIBU009158
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Diabetes Mellitus Nos New Onset; Hypertrophy, Left Ventricular; Vascular Stiffness
Keywords: Glucose Regulation; Left Ventricular Hypertrophy; New-onset Diabetes; Renal Transplantation
MeSH Terms: conditions — Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with New-onset Diabetes: New-onset diabetes after transplantation was defined as a fasting plasma glucose (FPG) level ≥ 126 mg/dL (7 mmol/L) or symptoms of diabetes plus casual plasma glucose concentrations ≥200 mg/dL (11.1 mmol/L), confirmed by repeat testing on a different day. According to these criteria, 63 patients were diagnosed as NODAT between years 2007-2010 but after the exclusion criteria of our study 57 patients with and 102 patients without NODAT were included in the study.
- Patients without NODAT: New-onset diabetes after transplantation was defined as a fasting plasma glucose (FPG) level ≥ 126 mg/dL (7 mmol/L) or symptoms of diabetes plus casual plasma glucose concentrations ≥200 mg/dL (11.1 mmol/L), confirmed by repeat testing on a different day. According to these criteria, 63 patients were diagnosed as NODAT between years 2007-2010 but after the exclusion criteria of our study 57 patients with and 102 patients without NODAT were included in the study.

SUMMARY:
New-onset diabetes (NODAT) after solid organ transplantation is an important clinical challenge associated to increased risk of cardiovascular (CV) events. In end-stage renal disease (ESRD) patients, the impact of arterial stiffness on all-cause and CV mortality has been clearly documented. Arterial stiffness has a pivotal role in the genesis of high blood pressure (SBP), increased left ventricular hypertrophy (LVH), and consequently CV mortality. Both LVH and arterial stiffness are independent determinants of CV disease in patients with ESRD. The aim of this study is to evaluate the relationship between post-transplant new-onset diabetes and arterial stiffness and left ventricular mass index (LVMI) in kidney transplant recipients.

DETAILED DESCRIPTION:
All patients' data were recorded from clinical charts. Visits in out patient clinic were organized as follows: three visits per week during the first 2 weeks; two visits per week until day 60; weekly visits until day 120; monthly visits during the first year; one visit every other month during the second year; and four visits per year thereafter until death or end-stage renal disease (i.e. dialysis or retransplantation). The following parameters were collected; 1) age, 2) gender, 3) posttransplantation duration, 4) pretransplant hemodialysis duration, 4) acute rejection episodes, 5) use of statins, ace inhibitor (ACE) or angiotensin receptor blocker (ARB), 6) immunosuppressive treatment (mycophenolate, cyclosporine, tacrolimus, and sirolimus use), 7) pretransplant lipid profile (values in the last month before transplantation), 8) posttransplant lipid profile (mean value), 9) FPG and HbA1c levels (mean value), 10) office blood pressure measurements, 11) hemoglobin, calcium, phosphorus, albumine and parathyroid hormone levels, 12) creatinine and estimated GFR (MDRD equation) and, 13) cytomegalovirus (CMV) infection history. Mean values were arithmetic means of each parameter that were collected from patient charts at 3 monthly basis after the first posttransplant 6 months while other parameters (12-16) were collected as single values at study inclusion.

All patients were under 5 mg prednisolone treatment within the immuno suppressive regimen. Maintenance immunosuppressive treatment included prednisone with a gradual tapering and mycophenolate mofetil or sodium associated with cyclosporine, tacrolimus or sirolimus in most patients. Target through levels at 3 months were 150-250 ng/ml for cyclosporine and 8-12 ng/ml for tacrolimus and sirolimus. Anti-diabetic treatment modalities (diet and lifestyle changes, oral anti-diabetic drugs or insulin) were also recorded for patients with NODAT.

Body compositions of all patients were analyzed by using the Body Composition Analyzer (Tanita BC-420MA). Fat mass, fat free mass, muscle mass, visceral fat mass and body mass index were calculated for each patient.

All patients underwent echocardiographic examinations (Siemens Acuson C256, Mountain view, California 2000 with 3V2c transducer probe) by the same operator and left ventricular mass was calculated according to the Devereux formula and indexed to body surface area to give LVMI (g/m2). Left ventricular mass index values greater than 130g/m2 (n: 57) were defined as high left ventricular mass.

Pulse wave velocity (PWv) is defined as the velocity of the arterial pulse for moving along the vessel wall. Pulse wave velocity along the aorta was measured by using two ultrasound or pressure sensitive transducers fixed transcutaneously over the course of a pair of arteries separated by a known distance: the femoral and right common carotid arteries. PWV was calculated from measurements of pulse transit time and the distance, according to the following formula: PWV (m/s)= distance (m)/transit time (s). Measurement of PWV values was con-ducted after abstinence from caffeine or smoking and after an overnight fast without intake of antihypertensive drugs. PWV was determined by using the SphygmoCor CvMs V9 system and values > 7 m/s was defined as increased.

ELIGIBILITY:
Inclusion Criteria:

Patients who underwent renal transplantation between years 2007-2010 in our transplantation clinic with routine periodical follow-up.

Exclusion Criteria:

* irregular drug usage or patient incompliance
* lack of regular follow-up data
* pretransplant diabetes mellitus history
* bone marrow transplant or other solid organs before or at the time of transplantation (including previous kidney transplantation)
* malign disease, rheumatologic or chronic inflammatory disease of unknown origin, systemic vasculitis history
* acute rejection periods after the first year of transplantation
* unstable cardiac disease including heart failure (ejection fraction < %50) and/or ischemic heart disease history (myocardial infarction, need for cardiac revascularization)
* atrial fibrillation or elevated heart rate (>100 beats/min)
* coronary bypass before or after transplantation
* transiently elevated fasting plasma glucose (FPG) or diabetic blood glucose profile during the first 3 posttransplant months
* graft failure [glomerular filtration (GFR) rate < 30 mL/min]
* history of peritoneal dialysis before transplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between years 2007-2010, 63 patients were diagnosed as NODAT in our transplantation center from the total 267 patients who underwent renal transplantation. Among these, 159 kidney transplant recipients were selected.
Sampling Method: Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Left ventricular hypertrophy | 3 years follow-up after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Siren Sezer, Prof. Dr., Study Chair — Baskent University, Department of Nephrology
Locations (1):
- Baskent University Medical School, Ankara, Turkey (Türkiye)